CLINICAL TRIAL: NCT00995644
Title: Natural History of Attempts to Stop Smoking
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Hughes, Professor of Psychiatry, University of Vermont
Other Study IDs: CHRBS #08-199; R01DA025089 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Tobacco Use Cessation
Keywords: smoking; smoking cessation; tobacco use cessation; tobacco use disorder
MeSH Terms: conditions — Tobacco Use Cessation; Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Smoking cessation can be enhanced either by increasing the success of quit attempts or by increasing in the number of quit attempts. The investigators are interested in what causes a smoker to make a quit attempt. The investigators will test whether certain events (e.g., a request from a child to quit smoking or exposure to a smoking-related health message) increase the probability of a quit attempt in the near future. The investigators are will test whether planning behaviors (e.g. seeking information about treatment) and setting a quit date are common and increase the probability of a quit attempt. Finally, the investigators want to see if spontaneous, unplanned quit attempts are common and are more or less successful than delayed, planned quit attempts. In a pilot study, the investigators will develop measures of the most common events and planning activities. In the main study, the investigators will recruit 200 adult daily smokers who are interested in quitting in the next 3 months. They will call a phone daily and use the phone's keypad to enter data plus they will complete mailed or internet questionnaires weekly for 3 months. The results of this study will a) help us understand what prompts smoking cessation attempts, b) help develop media messages and individual interventions to motivate smokers to make a quit attempt, and c) help determine whether spontaneous, impulsive quit attempts or delayed, planned quit attempts should be encouraged.

DETAILED DESCRIPTION:
METHODS Pilot Studies

One of our foci was on whether certain external events (prompts or cues) increase the probability of a quit attempt. We could not locate validated measures of possible external cues or planning activities for a quit attempt; thus, in Pilot Study 1, we recruited 28 daily, adult smokers of who had stopped smoking for at least 24 hours in the past month (including Hispanics, African-Americans, smokers whose income was below 1.5x poverty level, who were under age 24, and both men and women) to respond to a semi-structured telephone interview to identify possible causes of and preparations for their recent quit attempt. We used these responses to produce a list of 13 possible prompting events and two possible planning activities. In Pilot Study 2, we tested the ease of use of our IVR system and the clarity of our prompts. We will recruited smokers in the protocol described below including some who had a high school education or less and some who were 60 years or older. The only differences between this pilot study and the main study were that: a) IVR response options included a "don't know/unclear" option, and b) we will conduct a qualitative interview two weeks into the pilot 2 study to determine problems with IVR usage and understanding of the cue items. The pilot studies and the main study were approved by the University of Vermont Committees on the Use of Human Subjects.

Overview of Main Study

We will conduct a prospective cohort study of 200 adult daily smokers who were interested in quitting smoking in the next two months. Participants will call an interactive voice response (IVR) system daily for 3 months to report daily smoking, prompts to quit, planning events, and intentions to quit. In addition, they will complete more lengthy monthly questionnaires via mail or internet and, if they attempted to quit, a post-quit qualitative interview. We provided no intervention. The main aim was to determine which, if any, external cues to stop smoking or preparations for quitting prospectively increased the probability of a quit attempt. A secondary aim is to compare the predictive power of certain cessation-related internal cognitive variables versus external cues on quit attempts.

Participants

Participants will be recruited via newspaper and radio advertisements and via internet ads that will have messages such as "Daily cigarette smokers who plan to quit wanted for University of Vermont research study. Reimbursement for completing phone questions and mailed surveys. No need to leave home. This study does not offer treatment."

We chose a sample size of 200 because we believed about 50% of our sample would attempt to quit during the study period. This would provide 100 quit attempts which should be sufficient for prediction analyses. Plus a sample size of 200 produces a 95% confidence interval (CI) of no wider than + 7% with dichotomous outcomes.

Measures Participants will be given the option of completing baseline and monthly questionnaires either via return of mailed questionnaires or via a password-protected internet site. The baseline questionnaire will collect demographic and smoking information including past quit attempts, plans for quitting, and the Fagerstrom Test for Nicotine Dependence. It will ask the Mental Health Inventory (MHI), to indicate psychiatric problems and asked questions on recent alcohol and marijuana use and abuse.

Participants will complete the IVR questions nightly for 3 months. The IVR is a system in which participants call a number which directs them to enter data using the phone keypad. IVR has many of the assets of computer-assisted telephone interviewing; e.g., automatic skips, branching options, prohibition of illogical responses and outliers, standardized questioning, and direct data entry. IVR's major assets are the increased confidentiality, the ability to prompt participants to call, and the ability of participants to determine when to call. Drug use outcomes are more validly reported in IVR studies compared to in-person phone interviews, computer assessments, written questionnaires or in-person interviews. After brief training in the use of the IVR, participants will be instructed to call the IVR within 2 hours of their usual bedtime. If no call iss received during that window, the IVR telephoned the participant reminding them to call. The IVR questions include an assessment of current smoking status and whether the smoker plans to smoke tomorrow. If the participant reports smoking or being abstinent for only 1 day, the IVR asks whether each of 13 possible quit attempt cues and two planning activities (see Table 1) occurred on that day. If the participant reports abstinence for 2 or more days, the IVR will ask 12 questions about withdrawal symptoms and relapse cues, and whether abstinence was due to an attempt to stop smoking. If it was a quit attempt, a semi-structured interview will be scheduled to gain further details about the quit attempt and it's precipitants. To detect quit attempts that may not have lasted a full day, once each week the IVR will ask whether participants made a quit attempt that lasted less than a day in the past week.

At baseline and monthly, participants will complete questionnaires that ask about several cognitive variables related to stopping smoking; i.e., self-efficacy, perceived risks and benefits of smoking and abstinence and smoking expectancies.

Our major dependent variables are the events and cognitions and our major independent variable was the incidence of a quit attempt, defined as 24 hrs of abstinence due to an attempt to stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs of age
* smoke cigarettes daily for at least 1 year
* is able to read and write English
* as a final test of eligibility the investigators will determine if the person is compliant enough to participate in this study. The investigators will use 2 criteria:

  * they must complete 5 of 7 IVR sessions in the first week
  * they must complete the baseline questionnaires within one week of beginning the IVR sessions.

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
prediction of quit attempts | 3 mo

SECONDARY OUTCOMES:
success of quit attempts | 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hughes JR, Solomon LJ, Fingar JR, Naud S, Helzer JE, Callas PW. The natural history of efforts to stop smoking: a prospective cohort study. Drug Alcohol Depend. 2013 Feb 1;128(1-2):171-4. doi: 10.1016/j.drugalcdep.2012.08.010. Epub 2012 Aug 30. PMID 22939878
- [Result] Hughes JR, Solomon LJ, Naud S, Fingar JR, Helzer JE, Callas PW. Natural history of attempts to stop smoking. Nicotine Tob Res. 2014 Sep;16(9):1190-8. doi: 10.1093/ntr/ntu052. Epub 2014 Apr 9. PMID 24719491
- [Result] Hughes JR, Naud S, Fingar JR, Callas PW, Solomon LJ. Do environmental cues prompt attempts to stop smoking? A prospective natural history study. Drug Alcohol Depend. 2015 Sep 1;154:146-51. doi: 10.1016/j.drugalcdep.2015.06.044. Epub 2015 Jul 10. PMID 26190558